CLINICAL TRIAL: NCT00002019
Title: Safety and Efficacy of Amphotericin B Lipid Complex in the Treatment of Cryptococcal Meningitis in Patients With the Acquired Immunodeficiency Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liposome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 051A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-11

CONDITIONS: Meningitis, Cryptococcal; HIV Infections
Keywords: Meningitis; Liposomes; Cryptococcosis; Acquired Immunodeficiency Syndrome; Amphotericin B; Chemistry, Pharmaceutical
MeSH Terms: conditions — Meningitis, Cryptococcal; HIV Infections; Meningitis; Cryptococcosis; Acquired Immunodeficiency Syndrome | interventions — Amphotericin B

INTERVENTIONS:
Drug: Amphotericin B, Lipid-based
Drug: Amphotericin B

SUMMARY:
To evaluate the safety, tolerance and efficacy of three different dosage regimens of Amphotericin B Lipid Complex (ABLC) compared to Fungizone (Amphotericin B) in patients with AIDS and cryptococcal meningitis.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Intravenous pentamidine for treatment of Pneumocystis carinii pneumonia (PCP) but not for prophylaxis.

Patients must have the following:

* Meet the CDC criteria for diagnosis of AIDS.
* Confirmed episode of acute cryptococcal meningitis.
* Informed consent of the patient or guardian prior to entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Clinical evidence of acute or chronic meningitis due to an agent other than Cryptococcus neoformans.
* History of hypersensitivity/anaphylactoid reaction attributed to amphotericin B.
* Any other concomitant condition which, in the opinion of the investigator, would preclude a patient's participation in the study.

Concurrent Medication:

Excluded:

* Corticosteroids.
* Salicylates or other drugs known to interfere with prostaglandin synthesis except as specified in protocol.
* Zidovudine.
* Investigational agents.
* Interferon.
* Interleukin-2 (IL-2).
* Steroids.
* Isoprinosine.
* Intrathecal Amphotericin B.
* Intravenous Pentamidine PCP prophylaxis (only treatment).

Patients with the following are excluded:

* Clinical evidence of acute or chronic meningitis due to an agent other than Cryptococcus neoformans.
* History of hypersensitivity/anaphylactoid reaction attributed to amphotericin B.
* Inability to obtain appropriate follow-up visits.
* Any other concomitant condition which, in the opinion of the investigator, would preclude a patient's participation in the study.

Prior Medication:

Excluded within 4 weeks of study entry:

* Amphotericin B.
* Excluded within 2 weeks of study entry:
* Any other experimental drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Harbor - UCLA Med Ctr, Torrance, California
  - Dr Thomas Patterson, New Haven, Connecticut
  - Walter Reed Army Med Ctr, Washington D.C., District of Columbia
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Natl Naval Med Ctr, Bethesda, Maryland
  - Univ Hosp, Boston, Massachusetts
  - East Orange Veterans Administration Med Ctr, East Orange, New Jersey
  - Saint Michael's Med Ctr, Newark, New Jersey
  - Beth Israel Med Ctr / Peter Krueger Clinic, New York, New York
  - Dr Dorothy Friedberg, New York, New York
  - New York Univ Med Ctr, New York, New York
  - Cornell Univ Med College, New York, New York
  - Saint Luke's - Roosevelt Hosp Ctr, New York, New York
  - Mount Sinai Med Ctr / Jack Martin Fund Clinic, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Buckley Braffman Stern Med Associates, Philadelphia, Pennsylvania
  - Univ TX Galveston Med Branch, Galveston, Texas
  - Audie L Murphy Veterans Administration Hosp, San Antonio, Texas
  - Univ of Utah School of Medicine, Salt Lake City, Utah

REFERENCES:
- [Background] al-Haddadin D, Fan-Havard P, Boghossian J, Marton R, Vincent-Graber D, Dungo L, Eng RH, Johnson ES. Amphotericin B-lipid complex (ABLC) in treatment of cryptococcal meningitis in AIDS. Int Conf AIDS. 1992 Jul 19-24;8(2):B109 (abstract no PoB 3132)